CLINICAL TRIAL: NCT05105048
Title: A Phase 1, Randomized, Observer-Blind, Placebo-Controlled Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Cytomegalovirus Vaccine mRNA-1647 When Administered to Healthy Japanese Adults (18-40 Years of Age) in the United States
Brief Title: A Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Cytomegalovirus (CMV) Vaccine mRNA-1647
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1647-P103
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Cytomegalovirus Infection
Keywords: Moderna; mRNA-1647; Cytomegalovirus; CMV; Cytomegalovirus Vaccine; Cytomegalovirus Infections; Cytomegalovirus Congenital; Virus Diseases; Infection Viral; Messenger RNA
MeSH Terms: conditions — Cytomegalovirus Infections; Virus Diseases | interventions — mRNA-1647 cytomegalovirus vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1647 (Experimental): CMV-seronegative or CMV-seropositive participants will receive mRNA-1647 vaccine by intramuscular (IM) injection in a 0-, 2-, and 6-month schedule.
  Interventions: Biological: mRNA-1647
- Placebo (Placebo Comparator): CMV-seronegative or CMV-seropositive participants will receive placebo matching to mRNA-1647 vaccine by IM injection in a 0-, 2-, and 6-month schedule.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1647 — Lyophilized product that is reconstituted with saline
  Arms: mRNA-1647
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo

SUMMARY:
The main objective of this study is to evaluate the safety, reactogenicity, and immunogenicity of the mRNA-1647 vaccine administered according to a 3-study injection schedule in healthy cytomegalovirus (CMV)-seronegative and CMV-seropositive Japanese adults 18 to 40 years of age in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a Japanese Adult 18-40 years of age at the time of consent who, in the opinion of the investigator, is in good health based on review of medical history and screening physical examination. Japanese participants are defined as individuals born in Japan, with both parents and 4 grandparents who were born in Japan, and who have not lived outside of Japan for more than 10 years in total.
* For the CMV-seronegative groups: Participant is serum CMV IgG negative/ IgM negative.
* For the CMV-seropositive groups: Participant is either serum CMV IgG positive/IgM negative or IgG positive/IgM positive.
* Participant has a body mass index (BMI) from ≥18 kilograms (kg)/square meter (m^2) to ≤35 kg/m^2, inclusive.

Exclusion Criteria:

* History of a diagnosis or condition that, in the judgment of the investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures. Clinically unstable is defined as a diagnosis or condition requiring significant changes in management or medication within the 2 months prior to screening and includes ongoing workup of an undiagnosed illness that could lead to a new diagnosis or condition.
* Participant has elevated liver function tests, defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP), or elevated creatinine or reduced platelets, with a toxicity score of Grade ≥1 at screening.
* Participant has laboratory test results (hematology, chemistry, and coagulation) with a toxicity score of Grade ≥1 at screening.
* Received or plans to receive any non-study vaccine <28 days prior to any study injection; in addition, the following criteria for COVID-19 and influenza vaccines apply:

  i. Any COVID-19 vaccination series must have been completed a minimum of 28 days prior to receiving any dose of the study injection.

ii. COVID-19 vaccines (regardless of manufacturer) must be administered at least 28 days prior to or after any study injection.

iii. Influenza vaccines may be administered >14 days prior to or after any study injection.

* Participant has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months before the day of first injection (Day 1) (for corticosteroids, >5 mg/day of prednisone equivalent) or plans to do so during the course of the study. Inhaled, nasal, and topical steroids are allowed.
* Participant has received an antiviral with activity against CMV (ganciclovir, valganciclovir, foscarnet, cidofovir, letermovir, acyclovir, valacyclovir) within 2 weeks before the first injection or plans to do so during the course of the study.
* Participant received any investigational CMV vaccine.
* History of myocarditis, pericarditis, or myopericarditis.
* Reported medical history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV); or a positive screening test for hepatitis B surface antigen (HbSAg), hepatitis C antibodies, or HIV 1 or 2 antibodies.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 176 (7 days after each injection)
Number of Participants With Unsolicited Adverse Events (AEs) | Up to Day 197 (28 days after each injection)
Number of Participants With Medically-Attended AEs (MAAEs) | Day 1 through 6 months after the last injection (up to Day 347)
Number of Participants With Serious AEs (SAEs) | Day 1 through End of Study (EOS) (up to Day 347)
Number of Participants With AEs of Special Interest (AESIs) | Day 1 through EOS (up to Day 347)

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of Serum Neutralizing Anti-CMV Antibodies (nAbs) Against Epithelial Cell Infection and Against Fibroblast Infection | Days 1, 29, 85, 169, 197, and 347
Geometric Mean Fold-Rise (GMFR) of nAb Against Epithelial Cell Infection and Against Fibroblast Infection | Days 29, 85, 169, 197, and 347
Proportion of Participants with ≥2-Fold, 3-Fold, and 4-Fold Increases in nAb over Baseline Against Epithelial Cell Infection and Against Fibroblast Infection | Days 29, 85, 169, 197, and 347
GMT of Anti-Glycoprotein B (gB) Specific Immunoglobulin G (IgG) and Anti-Pentamer Specific IgG as Measured by Enzyme-Linked Immunosorbent Assay (ELISA) | Days 1, 29, 85, 169, 197, and 347
GMFR of Anti-gB and Anti-Pentamer Specific IgG | Days 29, 85, 169, 197, and 347
Proportion of Participants with ≥2-Fold, 3-Fold, and 4-Fold Increases Over Baseline in Anti-gB and Anti-Pentamer Specific IgG | Days 29, 85, 169, 197, and 347

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Velocity Clinical Research, North Hollywood, California
  - California Research Foundation, San Diego, California
  - East-West Medical Research Institute, Honolulu, Hawaii